CLINICAL TRIAL: NCT06760884
Title: Determination of Temporomandibular Joint Function, Oral Habits and Pain Complaints of Pregnant Women: a Cross-Sectional Case-Control Study
Brief Title: Temporomandibular Joint Function, Oral Habits and Pain Complaints of Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Principal Investigator, Karadeniz Technical University
Other Study IDs: KTU-FTR-2024/123
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Disorders (TMD); Pregnancy
Keywords: temporomandibular disorders; pregnancy; oral habits; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Pregnancy women
- Control group: Non-Pregnancy women

SUMMARY:
The aim of this study is to examine the temporomandibular joint functions, oral habits and pain complaints of pregnant women. .

DETAILED DESCRIPTION:
When looking at the literature, it is seen that physiological and hormonal changes that occur in pregnant women affect the musculoskeletal system and pain threshold of women. These changes seen in pregnant women and their psychological levels throughout the process also contribute negatively to the process.Due to the insufficiency of studies examining temporomandibular joint (TMJ) problems and oral habits in pregnant women and the contradictory results in existing studies, it is seen that new studies are needed.

ELIGIBILITY:
Inclusion Criteria (Pregnancy women):

* Being between the ages of 18-45,
* At least primary school graduate,
* Able to speak and understand Turkish,
* Women diagnosed with pregnancy by USG,
* Singleton pregnancy,
* Agreeing to participate in the study voluntarily.

Exclusion Criteria (Pregnancy women):

* Those with any systemic disease concerning the musculoskeletal system,
* Women with any type of disability,
* Having communication problems,
* Multiple pregnancy,
* Refusing to participate in the study.

Inclusion Criteria (Non-Pregnancy women):

* Being between the ages of 18-45,
* At least primary school graduate,
* Able to speak and understand Turkish,
* Agreeing to participate in the study voluntarily.

Exclusion Criteria (Non-Pregnancy women):

* Those with any systemic disease concerning the musculoskeletal system,
* Women with any type of disability,
* Having communication problems,
* Refusing to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females
Study Population: The universe of the study consists of women who apply to the pregnancy clinic. In parallel, a control group of 112 healthy non-pregnant women (similar to the pregnant group in terms of age, height, weight, education level, etc. to ensure homogeneity) will be created.
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Temporomandibular disorders function | 1 year
  Fonseca Anamnestic Index, which is reported as a reliable and valid index, will be used to evaluate the presence/absence of temporomandibular disorder and the severity of the disorder.
Mandibular function | 1 year
  The Mandibular Function Impairment Questionnaire (MFBA), a questionnaire that evaluates jaw function impairment with different sub-dimensions, will also be used.

SECONDARY OUTCOMES:
Oral Habits | 1 year
  The Oral Habits Checklist will be used.
Pain assessment | 1 year
  The presence, frequency and duration (how long has it been present) and severity of jaw, neck, back and waist pain will be questioned. The severity of pain will be assessed using the Numerical Pain Scale. This scale rates pain from "0" ("no pain") to "10" ("worst pain imaginable")

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical Univerity, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No